CLINICAL TRIAL: NCT04265911
Title: ASP3772 Phase 1 Study: Single Ascending Dose Study in Japanese Healthy Male and Female Adults, and PPSV23-controlled, Randomized, Single Ascending Dose Study in Japanese Elderly Male and Female Subjects
Brief Title: Single Ascending Dose of ASP3772 Study in Japanese Healthy Male and Female Adults, and Single Ascending Dose Study of ASP3772 in Comparison With PPSV23 in Japanese Elderly Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affinivax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3772-CL-1011
Record Dates: First submitted 2020-02-09; First posted 2020-02-12 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers
Keywords: Pneumococcal vaccine; ASP3772
MeSH Terms: interventions — Injections, Subcutaneous; Injections, Intramuscular; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- ASP3772 (subcutaneous) in Adults (Experimental): Participants will receive a single dose of ASP3772 administered as an subcutaneous injection on Day 1 at one of three dose levels.
  Interventions: Biological: ASP3772 (subcutaneous)
- ASP3772 ((intramuscular) in Adults (Experimental): Participants will receive a single dose of ASP3772 administered as an intramuscular injection on Day 1 at one of three dose levels.
  Interventions: Biological: ASP3772 (intramuscular)
- ASP3772 (subcutaneous) in Elderly (Experimental): Participants will receive a single dose of ASP3772 administered as an subcutaneous injection on Day 1 at one of three dose levels.
  Interventions: Biological: ASP3772 (subcutaneous)
- ASP3772 (intramuscular) in Elderly (Experimental): Participants will receive a single dose of ASP3772 administered as an intramuscular injection on Day 1 at one of three dose levels
  Interventions: Biological: ASP3772 (intramuscular)
- PPSV23 (subcutaneous) in Elderly (Active Comparator): Participants will receive a single subcutaneous injection of the standard dose of PPSV23 on Day 1.
  Interventions: Biological: PPSV23 (subcutaneous)
- PPSV23 (intramuscular) in Elderly (Active Comparator): Participants will receive a single intramuscular injection of the standard dose of PPSV23 on Day 1.
  Interventions: Biological: PPSV23 (intramuscular)

INTERVENTIONS:
Biological: ASP3772 (subcutaneous) — Subcutaneous injection
  Arms: ASP3772 (subcutaneous) in Adults; ASP3772 (subcutaneous) in Elderly
Biological: ASP3772 (intramuscular) — Intramuscular injection
  Arms: ASP3772 ((intramuscular) in Adults; ASP3772 (intramuscular) in Elderly
Biological: PPSV23 (subcutaneous) — Subcutaneous injection
  Other Names: Pneumovax NP
  Arms: PPSV23 (subcutaneous) in Elderly
Biological: PPSV23 (intramuscular) — Intramuscular injection
  Other Names: Pneumovax NP
  Arms: PPSV23 (intramuscular) in Elderly

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of 3 different dose levels of ASP3772 administered subcutaneously or intramuscularly to Japanese healthy adults 20 to 49 years of age.

This study will also evaluate the safety and tolerability of 3 different dose levels of ASP3772 administered subcutaneously or intramuscularly, in comparison to the active comparator 23-valent pneumococcal polysaccharide vaccine (PPSV23) in Japanese elderly subjects 65 to 85 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Subject is a healthy male or female between 20 and 49 years of age inclusive, at informed consent.
* Group 2: Subject is a male or female between 65 and 85 years of age inclusive, at informed consent who is healthy or has chronic controlled, stable disease with no change in disease severity, medical therapy and no hospitalization history in last 12 weeks from informed consent as determined by medical history, physical examination, and laboratory data.
* Female subject of non-childbearing potential; male subject not able to father children or who is able to father children and willing to use a highly effective method of contraception.
* Subject agrees not to participate in another interventional study while participating in the present study.
* Subject has a body mass index (BMI) range of 17.6 to 26.4 kg/m^2 inclusive in Group 1 and 15.4 to 28.6 kg/m^2 inclusive in Group 2, and body weight at least 50 kg for male and 40 kg for female at screening.

Exclusion Criteria:

* Subject has had previous vaccination with any licensed or investigational pneumococcal vaccine at any time.
* Subject has a history of microbiologically-proven invasive disease caused by Streptococcus pneumoniae.
* Subject has an immune disorder(s) (including autoimmune disease), clinical conditions requiring immunosuppressive drugs and/or a close relative who has congenital immunodeficiency.
* Group 1: Subject has any illness that requires medication or treatment.
* Group 2: Subject has any evidence of unstable or active clinically significant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease, e.g., uncontrolled hypertension, uncontrolled diabetes, heart failure, uncontrolled chronic obstructive pulmonary disease, end-stage renal disease, malignancy which is active and requires treatment.
* Subject has any clinically significant history of allergic conditions including drug allergies, asthma or anaphylactic reactions, but excluding untreated asymptomatic seasonal allergies just before study vaccine administration.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies (anti-HCV) or antigens/antibodies to human immunodeficiency virus (HIV) type 1 and/or type 2 at screening.
* Subject has/had febrile illness or symptomatic of viral, bacterial (including upper respiratory infection) or fungal (excluding skin infection) infection within 7 days prior to day 1.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2020-11-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with treatment emergent adverse events (TEAEs) including serious AEs (SAEs), medically attended adverse events (MAAEs), potentially immune mediated medical conditions (PIMMCs) and new onset chronic diseases (NOCDs) | Up to Day 30
  An adverse event (AE) is any untoward medical occurrence in a subject administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment. TEAE is defined as an AE occurring after study immunization to the last visit (up to 30 days post-vaccination if the study is discontinued for an individual subject). An IP-related TEAE is defined as any TEAE with a causal relationship assessed as "yes" by the investigator or subinvestigator.
Percentage of participants with vital sign abnormalities and/or adverse events (AEs) | Up to Day 30
  Percentage of participants with potentially clinically significant vital sign values.
Percentage of participants reporting solicited local adverse reactions | Up to Day 7
  Local reactions include pain, tenderness, erythema/redness, swelling, and induration. The reaction will be graded with 4-range grade: 1 (mild) to 4 (potentially life-threatening).
Percentage of participants reporting solicited systemic adverse reactions | Up to Day 7
  Systemic reactions include nausea, vomiting, diarrhea, headache, fever, fatigue and myalgia and arthralgia. Vital signs up to 7 days postvaccination are collected as systemic reactions. The reaction will be graded with 4-range grade: 1 (mild) to 4 (potentially life-threatening).
Percentage of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to Day 30
  Percentage of participants with potentially clinically significant laboratory values.
Percentage of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to Day 30
  Percentage of participants with potentially clinically significant ECG values.
Percentage of participants with physical exam abnormalities and/or adverse events (AEs) | Up to Day 30
  Percentage of participants with potentially clinically significant physical exam values.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) for opsonophagocytic activity (OPA) for each serotype contained in ASP3772 | On Day 30
  OPA measure will be used to characterize the immunological response on Day 30 after administration of ASP3772.
GMT for OPA for each serotype contained in PPSV23 | On Day 30
  OPA measure will be used to characterize the immunological response on Day 30 after administration of PPSV23
Ratio of the OPA GMT (each ASP3772 dose level/PPSV23) | On Day 30
  OPA measure will be used to characterize the immunological response on Day 30 after administration of ASP3772 and PPSV23
Geometric mean concentration (GMC) for pneumococcal serotype-specific anticapsular polysaccharide immunoglobulin G (PS IgG) for each serotype contained in ASP3772 | On Day 30
  PS IgG measure will be used to characterize the immunological response on Day 30 after administration of ASP3772.
GMC for pneumococcal serotype-specific anticapsular PS IgG for each serotype contained in PPSV23 | On Day 30
  PS IgG measure measure will be used to characterize the immunological response on Day 30 after administration of PPSV23
Ratio of GMC for pneumococcal serotype-specific anticapsular PS IgG (each ASP3772 dose level/PPSV23) | On Day 30
  PS IgG measure will be used to characterize the immunological response on Day 30 after administration of ASP3772 and PPSV23.
Geometric mean fold rise (GMFR) in anticapsular PS IgG concentration on day 30 relative to pre-immunization contained in ASP3772 | On Day 30
  PS IgG measure will be used to characterize the immunological response on Day 30 after administration of ASP3772.
GMFR in anticapsular PS IgG concentration on day 30 relative to pre-immunization contained in PPSV23 | On Day 30
  PS IgG measure will be used to characterize the immunological response on Day 30 after administration of PPSV23
GMFR in OPA titer on day 30 relative to pre-immunization contained in ASP3772 | On Day 30
  OPA titer will be used to characterize the immunological response on Day 30 after administration of ASP3772.
GMFR in OPA titer on day 30 relative to pre-immunization contained in PPSV23 | On Day 30
  OPA titer will be used to characterize the immunological response on Day 30 after administration of PPSV23
Proportion of subjects with a ≥ 4-fold increase relative to baseline in pneumococcal serotype-specific anticapsular PS IgG concentration for each serotype contained in ASP3772 | On Day 30
  PS IgG measure will be used to characterize the immunological response on Day 30 after administration of ASP3772.
Proportion of subjects with a ≥ 4-fold increase relative to baseline in pneumococcal serotype-specific anticapsular PS IgG concentration for each serotype contained in PPSV23 | On Day 30
  PS IgG measure will be used to characterize the immunological response on Day 30 after administration of PPSV23
Proportion of subjects with a ≥ 4-fold increase relative to baseline in OPA titer for each serotype contained in ASP3772 | On Day 30
  OPA titer will be used to characterize the immunological response on Day 30 after administration of ASP3772.
Proportion of subjects with a ≥ 4-fold increase relative to baseline in OPA titer for each serotype contained in PPSV23 | On Day 30
  OPA titer will be used to characterize the immunological response on Day 30 after administration of PPSV23

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (1):
- JP81001, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial as it meets one or more of the exceptions described on www.clinicalstudydatarequest.com under "Sponsor Specific Details for Astellas."

REFERENCES:
- [Derived] Borys D, Smulders R, Haranaka M, Nakano T, Chichili GR, Ebara M, Hashimoto A, Iwahana M, Oizumi Y, Nanra J, Malley R, Sebastian S. Safety, reactogenicity, and immunogenicity of a novel 24-valent pneumococcal vaccine candidate in healthy, pneumococcal vaccine-naive Japanese adults: A phase 1 randomized dose-escalation trial. Vaccine. 2025 Jan 12;44:126545. doi: 10.1016/j.vaccine.2024.126545. Epub 2024 Nov 29. PMID 39612802